CLINICAL TRIAL: NCT07091292
Title: Exercise Intervention as Treatment for People Using Cannabis (ExIT-C)-a Randomized Controlled Trial to Investigate the Effectiveness of Aerobic Exercise on Cannabis Dependence and Use Disorder
Brief Title: Exercise Intervention as Treatment for People Using Cannabis (ExIT-C)
Acronym: ExIT-C
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW 25-122
Record Dates: First submitted 2025-07-07; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-04

CONDITIONS: Cannabis Abuse; Cannabis Dependence; Cannabis Use Disorder
Keywords: exercise; cannabis; cannabis use disorder; cannabis dependence; substance abuse
MeSH Terms: conditions — Marijuana Abuse; Motor Activity; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Treatment (ExIT) Group (Experimental)
  Interventions: Behavioral: Indoor Cycling
- Sham-exercise Control (SCN) Group (Sham Comparator)
  Interventions: Behavioral: Indoor Cycling

INTERVENTIONS:
Behavioral: Indoor Cycling — Indoor cycling at 60-70% HR reserve for 30 minutes.
  Arms: Exercise Intervention Treatment (ExIT) Group
Behavioral: Indoor Cycling — Indoor cycling at 20-30% HR reserve for 30 minutes.
  Arms: Sham-exercise Control (SCN) Group

SUMMARY:
In Hong Kong, although the total number of drug abusers is trending down in recent years, the number of cannabis users continues to surge. The misuse of cannabis, if left unattended, predisposes various degrees of dependence and use disorders, which could later on induce psychotic disorders and schizophrenia. Effective strategies combating cannabis dependence and cannabis use disorder (CUD) are therefore warranted.

Exercise presents as a low-cost and low-stigma alternative to traditional pharmacotherapy and psychotherapy in the treatment of substance use disorders, which also promotes physical well-being with virtually no side effects. While exercise has some success in treating use disorders of stimulants, alcohol, and tobacco, evidence of its effects on CUD remains scarce. Hence, the present study will be conducted to assess the effectiveness of a 12-week aerobic exercise training regimen on reducing cannabis dependence and the severity of CUD.

Participants with cannabis dependence will be randomly assigned to either the exercise or the control group. Participants assigned to the exercise group will partake in a 12-week aerobic exercise training program of vigorous-intensity using indoor bikes, whereas those assigned to the control group will perform sham exercise of very light-intensity on indoor bikes. The 12-week study is divided into three (3) 4-week phases:

1. Intensive Intervention - all participants will exercise twice a week under supervision.
2. Active Intervention - all participants will exercise once a week under supervision.
3. Passive Maintenance - no supervised exercise sessions will be provided. All participants will receive exercise reminders via weekly text messages.

Cannabis use-related, cognitive, and physical outcomes will be assessed every 4 weeks, whereas withdrawal symptoms will be assessed and urine quick test administered every week.

ELIGIBILITY:
Inclusion Criteria:

* Young adults of 18-40 years old
* Able to read and communicate in English and/or Chinese
* Able to give informed consent
* Using cannabis or marijuana as the primary psychoactive substance of abuse
* Suffering from cannabis addiction, defined by:

  i. Cannabis Dependence with an SDS score ≥ 3, or ii. Cannabis Use Disorder according to the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5), or iii. Cannabis Harmful Use or Dependence according to the International Statistical Classification of Diseases and Related Health Problems 10th Revision (ICD-10) or Clinical descriptions and diagnostic requirements for International Classification of Diseases 11th Revision (ICD-11) mental, behavioral, and neurodevelopmental disorders.

Exclusion Criteria:

* Age < 18 or > 40 years old
* Unable to read English or Chinese
* Unable to give informed consent
* Absolute and/or relative contraindications to exercise training as indicated by the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+) and the electronic Physical Activity Readiness Medical Examination (ePARmed-X+)
* Had been diagnosed with the following disorders, including:

  i. Neurodevelopmental Disorders DSM-5: Intellectual Disabilities, Communication Disorders, Specific Learning Disorder, Autism Spectrum Disorder and Motor Disorders ICD-11: Disorders of intellectual development (6A00), Developmental speech or language disorders (6A01), Autism spectrum disorder (6A02), Developmental learning disorder (6A03), Developmental motor coordination disorder (6A04), Stereotyped movement disorder (6A06), Primary tics or tic disorders (8A05.0) ii. Other DSM-5 defined Substance Use Disorder greater than mild in severity (i.e., severity score ≥ 2), except for tobacco or caffeine iii. Neurocognitive Disorders (DSM-5, or ICD-11 6D70-72 & 6D80-86)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Diagnosis of Cannabis Use Disorder (CUD) | At enrollment and 4, 8, and 12 weeks after enrollment
  Structured Clinical Interview for DSM-5 Disorders (SCID-5) is used to ascertain the diagnosis and severity of CUD
Psychological Dependence on Cannabis | At enrollment and 4, 8, and 12 weeks after enrollment
  Severity of Dependence Scale (SDS) is used to assess psychological dependence on cannabis

SECONDARY OUTCOMES:
Urine Toxicology Test | At enrollment and 1, 2, 3, 4, 5, 6, 7, 8, and 12 weeks after enrollment
  Drug of Abuse Urine Test Kits is used to ascertain recent use of cannabis and/or other substances
Cannabis Craving | At enrollment and 4, 8, and 12 weeks after enrollment
  Marijuana Craving Questionnaire - Short Form (MCQ-SF) is used to assess cannabis craving
Cannabis Problems | At enrollment and 4, 8, and 12 weeks after enrollment
  Cannabis Problems Questionnaire (CPQ) is used to assess cannabis-related problems
Cannabis Withdrawal | At enrollment and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 weeks after enrollment
  Cannabis Withdrawal Scale (CWS) is used to assess cannabis withdrawal symptoms
Self-Efficacy in Cannabis Use Reduction | At enrollment and 4, 8, and 12 weeks after enrollment
  Marijuana Reduction Strategies Self-Efficacy Scale (MRSSES) is used to assess self-efficacy in reducing cannabis use
Self-reported Substance Use History | At enrollment and 4, 8, and 12 weeks after enrollment
  The frequency and amount of cannabis and substance use in the past 30 days is recorded
Global Cognitive Function | At enrollment and 4, 8, and 12 weeks after enrollment
  Montreal Cognitive Assessment - HK version (MoCA-HK) is used to assess global cognitive function
Psychomotor Speed | At enrollment and 1, 2, 3, 4, 5, 6, 7, 8, and 12 weeks after enrollment
  Digit Symbol Substitution Test (DSST) is used to assess psychomotor speed
Body weight (in kg) | At enrollment and 4, 8, and 12 weeks after enrollment
Height (in cm) | At enrollment
Waist circumference (in cm) | At enrollment and 4, 8, and 12 weeks after enrollment
Cardiopulmonary Capacity | At enrollment and 4, 8, and 12 weeks after enrollment
  Maximal oxygen uptake (V̇O2max) is measured to assess cardiopulmonary capacity
Resting Energy Expenditure | At enrollment and 4, 8, and 12 weeks after enrollment
Self-reported Physical Activity Participation | At enrollment and 9, 10, 11, and 12 weeks after enrollment
  International Physical Activity Questionnaire - Short Form (IPAQ-SF) is used to record the 7-day physical activity participation

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No